CLINICAL TRIAL: NCT04499976
Title: Adjuvant Isonicotinic Acid Hydrazide (INH) With Misoprostol for Induction of Abortion in First-trimester Missed Miscarriage Among Women With One or More Previous Cesarean Deliveries.: A Randomized Controlled Trial
Brief Title: Isonicotinic Acid Hydrazide Pretreatment With Misoprostol Induction of Abortion in First-trimester Missed Miscarriage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aswu/353/3/19
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Abortion, Missed
MeSH Terms: conditions — Abortion, Missed | interventions — Isonicotinic Acids; Misoprostol

STUDY DESIGN:
Intervention Model Description: double blind randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INH (Experimental): 3 tablets of isonicotinic acid hydrazide 300 mg will be given as single daily dose, 900 mg per day for two days at home and the third dose will be given on admission to hospital on day 3 and will be followed by vaginal misoprostol 800 mcg every three hours up to maximum two doses.
  Interventions: Drug: Isonicotinic Acid; Drug: Misoprostol
- Placebo Comparator (Placebo Comparator): three tablets of placebo will be given as a single daily dose, for two days at home and will be admitted on day 3 and continue treatment with misoprostol 800 mcg every three hours up to maximum two doses
  Interventions: Drug: Placebo; Drug: Misoprostol

INTERVENTIONS:
Drug: Isonicotinic Acid — Drug: Isonicotinic Acid then misoprostol Drug: Isonicotinic Acid 300mg total dose 900 mg per day for 3 days
  Arms: INH
Drug: Placebo — Drug: placebo then misoprostol Drug: Placebo placebo for 3 days
  Arms: Placebo Comparator
Drug: Misoprostol — Drug: Misoprostol Misoprosrol 800mcg will be given to all patients for induction of abortion

SUMMARY:
This study compares the success rate of Adjuvant isonicotinic acid hydrazide and misoprostol versus misoprostol alone for medical termination of first-trimester pregnancy among women with one or more previous cesarean deliveries.

DETAILED DESCRIPTION:
In the past, the role of laminaria and prostaglandins in cervical dilatation and reducing intraoperative complications of cervical dilatation have been proven . Misoprostol is a synthetic analogue of prostaglandin E1 used to treat and prevent gastric ulcers, which is now widely used in obstetrics and gynecology. Its applications in obstetrics and gynecology include medical abortion in the first and second trimesters of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than 70 days gestation (<10 wks).
* Hemoglobin >10 g/dL.
* BMI between 18.5 kg/m2 and 30 kg/m2.
* Missed abortion
* previous one or more cesarean deliveries

Exclusion Criteria:

* Molar pregnancy
* Fibroid uterus.
* Uterine anomalies.
* Coagulopathy
* Medical disorder that contraindicate induction of abortion (e.g. heart failure).
* Previous attempts for induction of abortion in the current pregnancy.
* Allergy to misoprostol or INH.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with one or more previous cesarean deliveries with missed miscarriage
Enrollment: 240 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
induction to abortion time | 9 hours
  induction to abortion time
number of patient with complete abortion | 9 hours
  number of patient with complete abortion

SECONDARY OUTCOMES:
number of patient need for surgical evacuation of the products of conception | 12 hours
  number of patient need for surgical evacuation of the products of conception

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No